CLINICAL TRIAL: NCT04876495
Title: Comparative Effects of Dairy and Plant-based Protein Intake on Acute Glucose Homeostasis and Appetite Regulation in Healthy Men
Brief Title: The Effects of Whey, Rice and Potato pRotein isOlates on appeTite rEgulatIoN in Healthy Men
Acronym: PROTEIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Westminster (Other)
Collaborators: Coventry University (Other)
Responsible Party: Principal Investigator, Mohammed Gulrez Zariwala, Professor of Translational Physiology, University of Westminster
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: VRE1516-1375
Record Dates: First submitted 2021-04-28; First posted 2021-05-06 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Appetite and General Nutritional Disorders
Keywords: nutraceutical; protein; whey; potato protein; rice protein; appetite; satiety; insulin; glucose; appetite hormone; GLP-1; PYY; supplement
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Intervention Model Description: single-blind, randomised, triple crossover
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Whey protein (Active Comparator): Whey protein isolate (45.5g total protein content)
  Interventions: Dietary Supplement: Whey protein isolate
- Potato protein (Active Comparator): Potato protein isolate (45.3g total protein content)
  Interventions: Dietary Supplement: Potato protein isolate
- Rice protein (Active Comparator): Rice protein isolate (45.5g total protein content)
  Interventions: Dietary Supplement: Rice protein isolate

INTERVENTIONS:
Dietary Supplement: Whey protein isolate — Instantized BiPRO® 50g (equiv. 45.5g of total protein) presented to participants in a form of a shake.
  Other ingredients in the whey protein shake:
  * Tropicana Trop50 Orange Juice 207mL
  * Water 43 mL
  * Sucralose 0.5g
  The total energy 233.47Kcal.
  Participants instructed to consume the entire protein shake presented to them in 5 minutes on an empty stomach when attending the study.
  Arms: Whey protein
Dietary Supplement: Potato protein isolate — Solanic®100 48g (equiv. 45.3g of total protein) presented to participants in a form of a shake.
  Other ingredients in the potato protein shake:
  * Tropicana Trop50 Orange Juice 250mL
  * Sucralose 0.5g
  The total energy 233.46Kcal
  Participants instructed to consume the entire protein shake presented to them in 5 minutes on an empty stomach when attending the study.
  Arms: Potato protein
Dietary Supplement: Rice protein isolate — Oryzatein® Silk 90 50g (equiv. 45.5g of total protein) presented to participants in a form of a shake.
  Other ingredients in the rice protein shake:
  * Tropicana Trop50 Orange Juice 183mL
  * Water 67mL
  * Sucralose 0.5g
  The total energy 233.43Kcal
  Participants instructed to consume the entire protein shake presented to them in 5 minutes on an empty stomach when attending the study.
  Arms: Rice protein

SUMMARY:
INTRODUCTION: Global protein consumption has been increasing for decades due to changes in socio-economic demographics and consumer trends towards higher protein intake, which may be related to their health benefits in performance nutrition and appetite regulation. The additional intake of protein often occurs in the form of supplements. One of the main ingredients used in sports and weight loss supplements are animal-derived proteins such as whey, which are of high quality, containing all the essential amino acids required in human nutrition with a high absorption rate. However, whey protein has a high environmental footprint, and it may contribute to insulin resistance in susceptible groups (e.g. obese, T2DM, insulin resistant, or those with sarcopenic obesity).

Rice and potato protein isolates are high-quality plant proteins containing all essential amino acids comparably to whey protein. These plant-derived proteins may provide a more sustainable and accessible alternative to animal-derived proteins for appetite regulation and weight management.

DETAILED DESCRIPTION:
Intervention study with three treatment groups in a randomised, single-blind, triple crossover design.

Study population: Healthy male participants will receive three different isocaloric and -volumetric protein shakes prepared using whey, rice and potato protein powders on different trial days with at least a one-week washout period apart.

Biological samples (blood and saliva samples) are collected at various time points during the visit. Blood samples are collected at baseline 10 min prior (T-10), then at 30 min (T30), 60 min (T60), 120 min (T120) and at 180 min (T180) after protein shake consumption. Saliva samples are collected at baseline (T-10), then at every 30 minutes following protein shake consumption (T30, T60, T90, T120, T150, T180). In addition, pertinent questionnaires Visual Analogue Scale [VAS] for the assessment of satiety and VAS for the assessment of protein shakes' perception will be collected at T-10, T30, T60, T90, T120, T150, T180 and at T0, respectively

ELIGIBILITY:
Inclusion Criteria:

* Males (18-65 years of age)
* Healthy subjects

Exclusion Criteria:

* <18 years or >65 years
* Consumption of >21 units of alcohol/week
* Dieters
* Any allergies/health issues related to items being ingested
* Any serious illnesses or those on medication
* Any illness affecting taste or appetite
* Any gastrointestinal disorders
* Any eating disorders
* Any depression/mental disorders
* Smoking

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants' eligibility is based on self-representation of gender identity
Enrollment: 12 (Actual)
Dates: Start 2018-07-20 (Actual); Primary Completion 2021-02-19 (Actual); Study Completion 2021-02-19 (Actual)

PRIMARY OUTCOMES:
To assess the acute effects of Solanic®100, Oryzatein® Silk 90 and Instantized BiPRO® on glucose levels (T-10) | Glucose measured 10 minutes prior to protein shake consumption
  Marker: glucose (mmol/L)
To assess the acute effects of Solanic®100, Oryzatein® Silk 90 and Instantized BiPRO® on glucose levels (T30) | Glucose measured 30 minutes post protein shake consumption
  Marker: glucose (mmol/L)
To assess the acute effects of Solanic®100, Oryzatein® Silk 90 and Instantized BiPRO® on glucose levels (T60) | Glucose measured 60 minutes post protein shake consumption
  Marker: glucose (mmol/L)
To assess the acute effects of Solanic®100, Oryzatein® Silk 90 and Instantized BiPRO® on glucose levels (T120) | Glucose measured 120 minutes post protein shake consumption
  Marker: glucose (mmol/L)
To assess the acute effects of Solanic®100, Oryzatein® Silk 90 and Instantized BiPRO® on glucose levels (T180) | Glucose measured 180 minutes post protein shake consumption
  Marker: glucose (mmol/L)
To assess the acute effects of Solanic®100, Oryzatein® Silk 90 and Instantized BiPRO® on insulin levels (T-10) | Insulin measured 10 minutes prior to protein shake consumption
  Marker: insulin (ng/mL)
To assess the acute effects of Solanic®100, Oryzatein® Silk 90 and Instantized BiPRO® on insulin levels (T30) | Insulin measured 30 minutes post protein shake consumption
  Marker: insulin (ng/mL)
To assess the acute effects of Solanic®100, Oryzatein® Silk 90 and Instantized BiPRO® on insulin levels (T60) | Insulin measured 60 minutes post protein shake consumption
  Marker: insulin (ng/mL)
To assess the acute effects of Solanic®100, Oryzatein® Silk 90 and Instantized BiPRO® on insulin levels (T120) | Insulin measured 120 minutes post protein shake consumption
  Marker: insulin (ng/mL)
To assess the acute effects of Solanic®100, Oryzatein® Silk 90 and Instantized BiPRO® on insulin levels (T180) | Insulin measured 180 minutes post protein shake consumption
  Marker: insulin (ng/mL)
To assess the acute effects of Solanic®100, Oryzatein® Silk 90 and Instantized BiPRO® on glucagon-like peptide 1 levels (T-10) | Glucagon-like peptide 1 measured 10 minutes prior to protein shake consumption
  Markers: glucagon-like peptide 1 (pM)
To assess the acute effects of Solanic®100, Oryzatein® Silk 90 and Instantized BiPRO® on glucagon-like peptide 1 levels (T30) | Glucagon-like peptide 1 measured 30 minutes post protein shake consumption
  Markers: glucagon-like peptide 1 (pM)
To assess the acute effects of Solanic®100, Oryzatein® Silk 90 and Instantized BiPRO® on glucagon-like peptide 1 levels (T60) | Glucagon-like peptide 1 measured 60 minutes post protein shake consumption
  Markers: glucagon-like peptide 1 (pM)
To assess the acute effects of Solanic®100, Oryzatein® Silk 90 and Instantized BiPRO® on glucagon-like peptide 1 levels (T120) | Glucagon-like peptide 1 measured 120 minutes post protein shake consumption
  Markers: glucagon-like peptide 1 (pM)
To assess the acute effects of Solanic®100, Oryzatein® Silk 90 and Instantized BiPRO® on glucagon-like peptide 1 levels (T180) | Glucagon-like peptide 1 measured 180 minutes post protein shake consumption
  Markers: glucagon-like peptide 1 (pM)
To assess the acute effects of Solanic®100, Oryzatein® Silk 90 and Instantized BiPRO® on peptide tyrosine tyrosine levels (T-10) | Peptide tyrosine tyrosine measured 10 minutes prior to protein shake consumption
  Markers: peptide tyrosine tyrosine (pg/mL)
To assess the acute effects of Solanic®100, Oryzatein® Silk 90 and Instantized BiPRO® on peptide tyrosine tyrosine levels (T30) | Peptide tyrosine tyrosine measured 30 minutes post protein shake consumption
  Markers: peptide tyrosine tyrosine (pg/mL)
To assess the acute effects of Solanic®100, Oryzatein® Silk 90 and Instantized BiPRO® on peptide tyrosine tyrosine levels (T60) | Peptide tyrosine tyrosine measured 60 minutes post protein shake consumption
  Markers: peptide tyrosine tyrosine (pg/mL)
To assess the acute effects of Solanic®100, Oryzatein® Silk 90 and Instantized BiPRO® on peptide tyrosine tyrosine levels (T120) | Peptide tyrosine tyrosine measured 120 minutes post protein shake consumption
  Markers: peptide tyrosine tyrosine (pg/mL)
To assess the acute effects of Solanic®100, Oryzatein® Silk 90 and Instantized BiPRO® on peptide tyrosine tyrosine levels (T180) | Peptide tyrosine tyrosine measured 180 minutes post protein shake consumption
  Markers: peptide tyrosine tyrosine (pg/mL)
To assess the acute effects of Solanic®100, Oryzatein® Silk 90 and Instantized BiPRO® on ghrelin levels (T-10) | Ghrelin (pg/mL) measured 10 minutes prior to protein shake consumption
  Markers: ghrelin (pg/mL)
To assess the acute effects of Solanic®100, Oryzatein® Silk 90 and Instantized BiPRO® on ghrelin levels (T30) | Ghrelin (pg/mL) measured 30 minutes post protein shake consumption
  Markers: ghrelin (pg/mL)
To assess the acute effects of Solanic®100, Oryzatein® Silk 90 and Instantized BiPRO® on ghrelin levels (T60) | Ghrelin (pg/mL) measured 60 minutes post protein shake consumption
  Markers: ghrelin (pg/mL)
To assess the acute effects of Solanic®100, Oryzatein® Silk 90 and Instantized BiPRO® on ghrelin levels (T120) | Ghrelin (pg/mL) measured 120 minutes post protein shake consumption
  Markers: ghrelin (pg/mL)
To assess the acute effects of Solanic®100, Oryzatein® Silk 90 and Instantized BiPRO® on ghrelin levels (T180) | Ghrelin (pg/mL) measured 180 minutes post protein shake consumption
  Markers: ghrelin (pg/mL)
To assess the acute effects of Solanic®100, Oryzatein® Silk 90 and Instantized BiPRO® on appetite (T-10) | Visual Analogue Scale for Appetite (VAS-A) collected immediately prior to protein shake consumption
  Subjective analysis including: Visual Analogue Scale for Appetite (VAS-A). Scores range from 0 to 100 (the higher the score the greater the level of appetite)
To assess the acute effects of Solanic®100, Oryzatein® Silk 90 and Instantized BiPRO® on appetite (T30) | Visual Analogue Scale for Appetite (VAS-A) collected 30 minutes after protein shake consumption
  Subjective analysis including: Visual Analogue Scale for Appetite (VAS-A). Scores range from 0 to 100 (the higher the score the greater the level of appetite)
To assess the acute effects of Solanic®100, Oryzatein® Silk 90 and Instantized BiPRO® on appetite (T60) | Visual Analogue Scale for Appetite (VAS-A) collected 60 minutes after protein shake consumption
  Subjective analysis including: Visual Analogue Scale for Appetite (VAS-A). Scores range from 0 to 100 (the higher the score the greater the level of appetite)
To assess the acute effects of Solanic®100, Oryzatein® Silk 90 and Instantized BiPRO® on appetite (T90) | Visual Analogue Scale for Appetite (VAS-A) collected 90 minutes after protein shake consumption
  Subjective analysis including: Visual Analogue Scale for Appetite (VAS-A). Scores range from 0 to 100 (the higher the score the greater the level of appetite)
To assess the acute effects of Solanic®100, Oryzatein® Silk 90 and Instantized BiPRO® on appetite (T120) | Visual Analogue Scale for Appetite (VAS-A) collected 120 minutes after protein shake consumption
  Subjective analysis including: Visual Analogue Scale for Appetite (VAS-A). Scores range from 0 to 100 (the higher the score the greater the level of appetite)
To assess the acute effects of Solanic®100, Oryzatein® Silk 90 and Instantized BiPRO® on appetite (T150) | Visual Analogue Scale for Appetite (VAS-A) collected 150 minutes after protein shake consumption
  Subjective analysis including: Visual Analogue Scale for Appetite (VAS-A). Scores range from 0 to 100 (the higher the score the greater the level of appetite)
To assess the acute effects of Solanic®100, Oryzatein® Silk 90 and Instantized BiPRO® on appetite (T180) | Visual Analogue Scale for Appetite (VAS-A) collected 180 minutes after protein shake consumption
  Subjective analysis including: Visual Analogue Scale for Appetite (VAS-A). Scores range from 0 to 100 (the higher the score the greater the level of appetite)

SECONDARY OUTCOMES:
To assess the perception of Solanic®100, Oryzatein® Silk 90 and Instantized BiPRO® | VAS for Palatability collected immediately after protein shake consumption
  Subjective analysis including: Visual Analogue Scale for Palatability (VAS-P). Scores range from 0 to 100 (the higher the score the lower the palatability)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Gulrez Zariwala, PhD, Principal Investigator — University of Westminster
Locations (1):
- University of Westminster, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: No